CLINICAL TRIAL: NCT02969460
Title: Neurotrack Virtual Cognitive Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: Neurotrack (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EH-003
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Subjective Cognitive Decline

ARMS (1):
- Neurotrack Virtual Cognitive Health Program (Experimental): This program is a multi-domain lifestyle intervention designed to prevent or delay cognitive decline and impairment in older at-risk adults. The first 6 months of the program emphasizes lifestyle change, while the last 6 months of the program emphasizes habit reinforcement. The program focuses on nutrition, physical exercise, and cognitive training.
  Interventions: Behavioral: Neurotrack Virtual Cognitive Health Program

INTERVENTIONS:
Behavioral: Neurotrack Virtual Cognitive Health Program

SUMMARY:
The Neurotrack Virtual Cognitive Health Study is a 12-month long, prospective study that aims to evaluate the impact of the Neurotrack Virtual Cognitive Health Coaching Program on cognitive ability, anxiety and depression, and lifestyle behaviors for individuals who show signs of subjective cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Ages 60-75
* Individuals who show signs of subjective cognitive decline (assessed by scoring ≥ 1 on the Subjective Cognitive Decline [Short Form] Questionnaire and endorsing the Personal Worry Item on the questionnaire)
* Have the ability to make and receive phone calls
* Have the ability to send and receive text messages
* Access to a desktop computer, video-teleconferencing and reliable internet connection
* Motivated to use a daily coaching program

Exclusion Criteria:

* Significant history of mental illness, substance abuse, learning disability, or neurologic conditions
* History of dementia
* Ophthalmologic/visual problems that prevent individual from viewing a computer screen at a normal distance (e.g., legal blindness, detached retinas, occlusive cataracts)
* Currently participating in a formal cognitive-training coaching program
* Currently pregnant

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
RBANS score | week 24
  Repeatable Battery for the Assessment of Neuropsychological Status total score
RBANS score | week 52
  Repeatable Battery for the Assessment of Neuropsychological Status total score

SECONDARY OUTCOMES:
PHQ-9 | week 24
  Patient-health questionnaire 9-item scale
PHQ-9 | week 52
  Patient-health questionnaire 9-item scale
GAD-7 | week 24
  Generalized anxiety disorder 7-item scale
GAD-7 | week 52
  Generalized anxiety disorder 7-item scale

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, San Mateo, California, United States

REFERENCES:
- [Derived] Kumar S, Tran J, Moseson H, Tai C, Glenn JM, Madero EN, Krebs C, Bott N, Juusola JL. The Impact of the Virtual Cognitive Health Program on the Cognition and Mental Health of Older Adults: Pre-Post 12-Month Pilot Study. JMIR Aging. 2018 Nov 9;1(2):e12031. doi: 10.2196/12031. PMID 31518248
- [Derived] Bott N, Kumar S, Krebs C, Glenn JM, Madero EN, Juusola JL. A Remote Intervention to Prevent or Delay Cognitive Impairment in Older Adults: Design, Recruitment, and Baseline Characteristics of the Virtual Cognitive Health (VC Health) Study. JMIR Res Protoc. 2018 Aug 13;7(8):e11368. doi: 10.2196/11368. PMID 30104186